CLINICAL TRIAL: NCT07179926
Title: Effects of Pasireotide Lar Therapy on Bone Metabolism
Acronym: Pasi-Bone
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7394
Record Dates: First submitted 2025-06-24; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Acromegaly Due to Pituitary Adenoma; Acromegaly
MeSH Terms: conditions — Growth Hormone-Secreting Pituitary Adenoma; Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PROSPECTIVE COHORT: PROSPECTIVE COHORT switched to Pasireotide LAR after fg-SRLs, according to clinical practice
  Interventions: Diagnostic Test: morphometric spine radiography
- RETROSPECTIVE COHORT: RETROSPECTIVE COHORT switched to Pegvisomant after fg-SRLs, according to clinical practice
  Interventions: Diagnostic Test: morphometric spine radiography

INTERVENTIONS:
Diagnostic Test: morphometric spine radiography — Patients already on treatment with Pasireotide LAR or Pegvisomant will be evaluated using morphometric spine radiography and lumbar and femoral densitometry. Patients will undergo a 1-year follow-up.
  Other Names: lumbar and femoral densitometry

SUMMARY:
Acromegaly, a chronic condition characterized by growth hormone (GH) and, in turn, insulin-like growth factor-1 (IGF-I) excess, is burdened by a series of systemic and metabolic comorbidities that strongly impair quality of life (QoL) and life expectancy. Amongst them, a specific acromegalic osteopathy has been discovered, characterized by fragility fractures associated with high bone turnover, which need to be early detected, according to most recent guidelines, since they are very frequent and related to chronic pain and reduced QoL. Morphometric vertebral fractures (VFs) are an emerging landmark of skeletal fragility in general population as well as in clinical trials, and are highly prevalent in acromegaly, being reported to affect from 30 up to 60% of patients and represent an early and common event in disease history. Until now, same groups of patients with higher risk of vertebral fractures were identified, such as those carrying incident vertebral fractures, or affected by biochemical active acromegaly, concomitant hypogonadism, or diabetes mellitus. The main aim in the management of patients with acromegaly is to normalize IGF-I levels and restore acromegaly related symptoms. To aim this treatment objective, the first line of treatment of acromegaly, when feasible, is neurosurgery. In cases where surgical intervention fails to achieve biochemical control, medical therapy is recommended, with the objective of reaching normal levels of IGF-1 and GH age-corrected. Octreotide LAR and Lanreotide are the first-line medical therapy. In patients who have not achieved adequate control with standard doses of octreotide LAR and Lanreotide, increasing the dose and/or frequency of administration can lead to improved biochemical control. In patients who are unable to achieve control even with this approach, a switch to Pasireotide LAR may be considered. In instances where patients fail to achieve biochemical control with maximal doses of SRL, or in the presence of contraindications, the use of Pegvisomant as a second-line therapy may be considered. In addition, a combination of Pegvisomant and SRL represents a potential avenue for treating patients. Prevention of VFs in acromegaly remains an open issue. It has been shown that use of GH/IGF-I lowering treatments with first-generation SSA and Pegvisomant, may reduce the risk of VFs, while improving disease control. Moreover, in a retrospective and observational multicenter study, it was recently proved that patients treated with second generation SRLs (Pasireotide-LAR) developed less frequently VFs then patients treated with Pegvisomant.

ELIGIBILITY:
INCLUSION CRITERIA FOR THE PROSPECTIVE COHORT

* adult patients (>18 years)
* acromegaly not-controlled after 6 months of treatment with fg-SRLs and switched since at least one week, to Pasireotide LAR, according to clinical practice and actual experts consensus,
* signing of informed consent

INCLUSION CRITERIA FOR THE RETROSPECTIVE COHORT

* adult patients (>18 years)
* acromegaly not-controlled after 6 months of treatment with fg-SRLs and switched to Pegvisomant, according to clinical practice and actual experts' consensus,
* signing of informed consent or substitute declaration on the consent form where applicable.

Exclusion Criteria:

* patients under the age of 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: n the prospective cohort will be included patients with diagnosis of acromegaly not-controlled after 6 months of treatment with first generation somatostatin receptor ligands (SRLs) with IGF-I upper the age-adjusted limit of normality, and treated for at least one week with Pasireotide Lar, according to clinical practice In the retrospective cohort will be included patients with diagnosis of acromegaly not-controlled after 6 months of treatment with first generation somatostatin receptor ligands (SRLs) with IGF-I upper the age-adjusted limit of normality, and treated with Pegvisomant from 01.01.2010 to 31-12- 2024 (including follow-up data).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Comparison between Pasireotide LAR and Pegvisomant | 36 months
  The primary objective is to evaluate the rate of incidental vertebral fractures over 12 consecutive months of treatment with Pasireotide LAR, in comparison to the historical control arm which received Pegvisomant monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Chiloiro, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS UOC Endocrinologia e Diabetologia, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No